CLINICAL TRIAL: NCT01241500
Title: Phase III MultiCenter Randomized Controlled Study to Assess Efficacy and Safety of ON 01910.Na 72-Hr Continuous IV Infusion in MDS Patients With Excess Blasts Relapsing After or Refractory to or Intolerant to Azacitidine or Decitabine
Brief Title: Randomized Study of ON 01910.Na in Refractory Myelodysplastic Syndrome Patients With Excess Blasts
Acronym: ONTIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-21
Record Dates: First submitted 2010-11-01; First posted 2010-11-16 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2018-07

CONDITIONS: Myelodysplastic Syndromes; MDS; RAEB; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic syndromes; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ON 01910.Na + best supportive care (BSC) (Experimental): Patients will receive ON 01910.Na 1800 mg/24 hr as a continuous intravenous infusion for 72 hours every other week for the first 16 weeks then every 4 weeks afterwards and best supportive care (BSC).
  Interventions: Drug: ON 01910.Na
- Best supportive care (BSC) (No Intervention): Patients will receive best supportive care (BSC).

INTERVENTIONS:
Drug: ON 01910.Na — The dose of ON 01910.Na will be 1800 mg/24 hr as a continuous intravenous infusion for 72 hours every other week for the first 16 weeks then every 4 weeks afterwards. Infusion bags must be changed every 24 hours and a new infusion bag must be used for each of the subsequent 24 hours until completion of the total 72-hour infusion time.
  Other Names: rigosertib
  Arms: ON 01910.Na + best supportive care (BSC)

SUMMARY:
The primary objective of this study is to compare overall survival (OS) in patients receiving ON 01910.Na + best supportive care (BSC) to OS of patients receiving BSC in a population of patients with myelodysplastic syndrome (MDS) with excess blasts (5% to 30% bone marrow blasts) who have failed azacitidine or decitabine treatment. This patient population has no available therapy and a short life expectancy (approximately 4 months). The high level of bone marrow activity of ON 01910.Na documented in Phase 1 and 2 studies has the potential to delay substantially the transition of MDS to Acute Myeloid Leukemia(AML), a very significant and severe complication, which shortens survival of these MDS patients.

DETAILED DESCRIPTION:
This is a Phase III open-label, randomized, controlled, multicenter study (up to 50 centers). Approximately 270 patients with MDS classified as RAEB-1 and RAEB-2 using the WHO classification and as RAEB-t and chronic myelomonocytic leukemia (CMML) using the FAB classification who failed, became intolerant to, or progressed after treatment with 5-azacitidine or decitabine administered during the past 2 years, will be randomized in a 2:1 ratio into the following 2 treatment regimens:

* Best Supportive Care (BSC) + ON 01910.Na 1800 mg/24 hr administered as a 72-hr continuous intravenous (CIV) infusion on Days 1, 2, and 3 of a 2-week cycle (N = approximately 180 patients)
* BSC (N = approximately 90 patients).

Patients will be stratified at entry by bone marrow (BM) blasts (5% to 19% vs. 20% to 30%). After completing the first eight 2-week cycles (i.e., after 16 weeks of treatment), the frequency of further 72-hr CIV infusions will be decreased to an administration on Days 1, 2, and 3 of a 4-week cycle.

Patients will remain treated on study until 2006 International Working Group (IWG) progression criteria are met (i.e., 50% increase of BM blasts or worsening of cytopenias) or until death from any cause, whichever comes first.

Patients who progress to Acute Myeloid Leukemia (AML) while on study should be offered either standard treatment for AML or enrollment in an appropriate investigational study if they are eligible. These treatments with their start and end dates should be documented and patient survival time will be documented for all randomized patients.

Cross-over of BSC patients to ON 01910.Na after progression will not be allowed. However, patients in the BSC-only group will be allowed, as medically justified, access to low-dose cytarabine 20 mg/m2 subcutaneously (SC) once daily for the first consecutive 14 days of each 28-day cycle, up to 4 cycles, until progression or unacceptable toxicity develops. Low-dose cytarabine will be delayed as needed until recovery of blood counts. All study participants will be allowed, as medically justified, access to RBC and platelet transfusions and to growth factors (erythropoietin, Filgrastim [G-CSF]). Hydroxyurea will be allowed to manage blastic crisis with hyperleukocytosis when patients transition to leukemia.

ELIGIBILITY:
Inclusion Criteria:

* MDS diagnosis confirmed within 6 weeks prior to entry according to WHO or FAB classification
* MDS classified as follows, according to WHO and FAB classification:

  * RAEB-1 (5% - 9% BM blasts)
  * RAEB-2 (10% - 19% BM blasts)
  * CMML (10% - 20% BM blasts) and WBC < 13,000/μL
  * RAEB-t (20% - 30% BM blasts), with following criteria:
  * o WBC < 25 x 10E9/L at entry
  * o Stable WBC at least 4 weeks prior to entry and not requiring intervention for WBC control with hydroxyurea, chemotherapy, or leukopheresis.
* At least one cytopenia (ANC < 1800/µL or platelet count < 100,000/µL or hemoglobin <10 g/dL)
* Progression according to 2006 International Working Group (IWG) criteria any time after start of azacitidine or decitabine during past 2 years; or failure to achieve complete or partial response or hematological improvement (according to 2006 IWG) after at least six 4-week cycles of azacitidine or four 6-week cycles of decitabine during past 2 years; or relapse after initial complete or partial response or hematological improvement (according to 2006 IWG criteria) observed after at least six 4-week cycles of azacitidine or four 6-week cycles of decitabine during past 2 years; or, intolerance to azacitidine or decitabine defined by drug-related ≥Grade 3 liver or renal toxicity leading to discontinuation during the past 2 years.
* Did not respond to, relapsed after, not eligible for, or opted not to do bone marrow transplantation
* Off other MDS treatments for at least 4 weeks; Filgrastim (G-CSF) and erythropoietin allowed before and during the study as clinically indicated.
* No need for induction chemotherapy
* ECOG status 0, 1 or 2
* Willing to adhere to protocol prohibitions and restrictions
* Patient (or a legally authorized representative) must sign informed consent form to indicate patient's understanding study's purpose and procedures and willingness to participate

Exclusion Criteria:

* Anemia due to factors other than MDS (including hemolysis or gastrointestinal bleeding) unless stabilized for 1 week after RBC transfusion.
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy
* Total bilirubin ≥1.5 mg/dL not related to hemolysis or Gilbert's disease.
* Alanine transaminase (ALT)/aspartate transaminase (AST) ≥2.5 x upper limit of normal (ULN)
* Serum creatinine ≥2.0 mg/dL
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 mEq/L)
* Pregnant or lactating females
* Patients unwilling to follow strict contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine device, double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) before entry and throughout the study
* Females with reproductive potential who do not have a negative urine beta-human chorionic gonadotropin pregnancy test at screening
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start
* Uncontrolled hypertension (defined as systolic pressure ≥160 mmHg and/or diastolic pressure ≥110 mmHg)
* New onset seizures (within 3 months prior to first dose of ON 01910.Na) or poorly controlled seizures
* Any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy
* Prior treatment with low-dose cytarabine during past 2 years Investigational therapy within 4 weeks of starting ON 01910.Na
* Psychiatric illness or social situation that limits the patient's ability to tolerate and/or comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 18 months
  Overall survival (OS) is defined as the time from randomization to death from any cause. All patients will be followed until death or progression, even if they have discontinued treatment for whatever cause. Patients lost to follow-up will be censored at the time last known alive. The OS primary analysis will compare the active ON 01910.Na regimen to BSC once a total number of 223 deaths has been reached.

SECONDARY OUTCOMES:
Overall response (complete and partial remission) according to 2006 IWG criteria | Changes measured at Week 4 from Baseline and every 8 Weeks thereafter
  Compare the BSC + ON 01910.Na group to the BSC group with respect to changes in bone marrow myeloblasts, hemoglobin, peripheral neutrophils, platelets and blasts.
Complete bone marrow response according to 2006 IWG criteria | Changes measured at Week 4 from Baseline and every 8 Weeks thereafter
  Compare the BSC + ON 01910.Na group to the BSC group with respect to changes in bone marrow myeloblasts.
Hematological improvements according to 2006 IWG criteria | Weekly
  Compare the BSC + ON 01910.Na group to the BSC group with respect to in absolute neutrophil count (ANC), platelet count, and erythroid responses.
Scores of Quality of Life Questionnaire | Measured at Baseline and every 4 Weeks
  Compare the BSC + ON 01910.Na group to the BSC group with respect to scores of Quality-of-life (QOL)(using the European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-C30 version 3.
Adverse events | Weekly
  Record adverse events according to CTCAE v4.
Change in Aneuploidy | Baseline and, only if abnormal at Baseline, Week 4 and every 8 Weeks thereafter
  Improvements of cytogenetics as evaluated by the change in aneuploidy in bone marrow according to 2006 IWG criteria.
Transition time to AML | Measured at Week 4 from date of randomization and every 8 Weeks thereafter
  Transition time to AML: Defined for RAEB-1 and RAEB-2 MDS and chronic myelomonocytic leukemia (CMML) patients (with BM blasts from 10% to 20% for CMML) by an increase of at least 50% BM blasts and more than 20% BM blasts; Defined for RAEB-t by an increase of at least 50% BM blasts.
Incidence of infections and bleeding episodes. | Every 4 Weeks
  Incidence of infections (treated with intravenous antimicrobials) and bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Chair — Traws Pharma, Inc.
Locations (87):
- United States (41):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Center, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Mount Sinai Comprehensive Cancer Centers, Miami Beach, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Martin Memorial Cancer Center, Stuart, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - North Shore Medical Center, Evanston, Illinois
  - Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - North Shore - LIJ Health System, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francois Health System, Greenville, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - H. Hartziekenhuis Roeselare-Menen vzw, Roeselare, West-vlaanderen
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - CHU de Mont-Godinne, Yvoir
- France (15):
  - CHU Angers Service de Medecine D - Maladies du Sang, Angers
  - CHU Avignon Centre Hospitalier Henri Dufaut, Avignon
  - Hôpital Avicenne Hématologie Clinique, Bobigny
  - CHU Caen Hématologie Clinique, Caen
  - CHU Estaing Service d'hématologie, Clermont-Ferrand
  - CHU Lille Hôpital Claude Huriez, Lille
  - CHU Limoges Hopital Dupuytren, Limoges
  - Institute Paoli Calmettes, Marseille
  - Hôpital de L'archet I, Nice
  - Hôtel Dieu Sce Hématologie Clinique, Paris
  - Hôpital Saint-Antoine, Paris
  - CHU Perpignan Centre Hospitalier Hôpital Saint-Jean, Perpignan
  - CRLCC Henri Becquerel, Rouen
  - Chu-Strasbourg-Hopital Civil, Strasbourg
  - Hôpital Purpan, Toulouse
- Germany (10):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum zu Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - Klinikum der Johann Wolfgang-Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsmedizin Mannheim, Mannheim
  - Johannes-Wesling-Klinikum Minden, Minden
  - Klinikum Rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Ulm, Ulm
- Italy (9):
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte, Siena, SI
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero-Universitaria di Bologa Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera-Universitairia Vittorio Emanuele-Ferrarotto-Santo Bambino, Catania
  - Azienda Ospedaliera Universitaria Careggi di Firenze, Florence
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Osperdaliera Universitaria Maggiore della Carità, Novara
  - Università degli Studi La Sapienza, Roma
  - Azienda Ospedaliero Universitaria San Giovanni Battista di Torino, Torino
- Spain (8):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Background] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Background] Athuluri-Divakar SK, Vasquez-Del Carpio R, Dutta K, Baker SJ, Cosenza SC, Basu I, Gupta YK, Reddy MV, Ueno L, Hart JR, Vogt PK, Mulholland D, Guha C, Aggarwal AK, Reddy EP. A Small Molecule RAS-Mimetic Disrupts RAS Association with Effector Proteins to Block Signaling. Cell. 2016 Apr 21;165(3):643-55. doi: 10.1016/j.cell.2016.03.045. PMID 27104980
- [Result] Garcia-Manero G, Fenaux P, Al-Kali A, Baer MR, Sekeres MA, Roboz GJ, Gaidano G, Scott BL, Greenberg P, Platzbecker U, Steensma DP, Kambhampati S, Kreuzer KA, Godley LA, Atallah E, Collins R Jr, Kantarjian H, Jabbour E, Wilhelm FE, Azarnia N, Silverman LR; ONTIME study investigators. Rigosertib versus best supportive care for patients with high-risk myelodysplastic syndromes after failure of hypomethylating drugs (ONTIME): a randomised, controlled, phase 3 trial. Lancet Oncol. 2016 Apr;17(4):496-508. doi: 10.1016/S1470-2045(16)00009-7. Epub 2016 Mar 9. PMID 26968357
- [Result] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Al-Kali A. Relationship of bone marrow blast (BMBL) response to overall survival (OS) in a multicenter study of rigosertib (Rigo) in patients (pts) with myelodysplastic syndrome (MDS) with excess blasts progressing on or after treatment with a hypomethylating agent (HMA). Journal of Clinical Oncology 2017 35:15_suppl, 7056-7056 ASCO 2017
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Leukemia and Lymphoma Society — http://www.lls.org/
- See also: The Myelodysplastic Syndromes Foundation — http://mds-foundation.org/